CLINICAL TRIAL: NCT04326777
Title: Balloon Pulmonary Angioplasty for Patients With Chronic Thromboembolic Pulmonary Hypertension: A Single-center, Prospective Long-term Follow-up Study
Brief Title: Clinical Study of Balloon Pulmonary Angioplasty for Patients With Chronic Thromboembolic Pulmonary Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Li Xuyan (Other)
Responsible Party: Sponsor-Investigator, Li Xuyan, Deputy Director of Respiratory and Critical Care Medicine,Beijing Institute of Respiratory Medicine, Beijing Chaoyang Hospital, Capital Medical University, Beijing Chao Yang Hospital
Organization: Beijing Chao Yang Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-KE-377
Record Dates: First submitted 2020-03-27; First posted 2020-03-30 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension
Keywords: Balloon pulmonary angioplasty(BPA); Chronic Thromboembolic Pulmonary Hypertension(CTEPH)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ballon pulmonary angioplasty (Other): Ballon pulmonary angioplasty(BPA) is a stepwise procedure requiring several separate sessions. The interval of a series of BPA is one month. In a series of BPA, there are 2 sessions, which are repeated at a 2-week interval. BPA is performed primarily on one side of the lung in the first session, then after 2 weeks, performed on the other side of the lung. In each session, the fluoroscopy time or the amount contrast are less than 60min and 200ml, respectively.
  Interventions: Procedure: Ballon pulmonary angioplasty

INTERVENTIONS:
Procedure: Ballon pulmonary angioplasty — Percutaneous vascular access for BPA is via the femoral vein using Seldinger technique. A 5Fr sheath is inserted into the vein, through which a 6Fr long introducer sheath is advanced into the pulmonary artery. Subsequently, a 6Fr guiding catheter is advanced into the pulmonary artery being treated. Generally, selective pulmonary angiography should be performed to evaluate lesion feature before BPA. Then a 0.014-inch guidewire is used to cross the lesion, a balloon catheter of an appropriate diameter is selected to dilate the lesion.

SUMMARY:
Chronic thromboembolic pulmonary hypertension (CTEPH) is the fourth group of pulmonary hypertension (PH) according to clinical classification. Pulmonary endarterectomy（PEA) is the preferred treatment for patients with CTEPH, however, PEA has its limitations, it only applies to the thrombi in the main, lobar, or segmental pulmonary arteries for patients with CTEPH, and the postoperative residual PH is found to be of high percentage. With the development of interventional techniques, balloon pulmonary angioplasty (BPA) has been used to treat chronic thrombotic pulmonary hypertension (CTEPH) with favorable results and has been identified as an effective and safe treatment for technically inoperable CTEPH. Balloon pulmonary angioplasty (BPA) has been accepted as a therapeutic strategy in accordance with the 2015 ESC/ESR guidelines, especially for patients with technically inoperable, an unfavorable risk-to-benefit ratio of the PEA. This study was a single-center prospective study that collects 3 time points data (before BPA, after final BPA, and follow-up ) to verify long-term safety and efficacy of BPA, as well as comparing the efficacy with targeted medical therapy, evaluating the complications of BPA, the survival of patients, and the postoperative quality of life.

ELIGIBILITY:
Inclusion Criteria:

* technically inoperable for PEA in patients with CTEPH
* unfavorable risk/benefit ratio for PEA
* residual or recurrent PH after PEA
* aged over 18 years old

Exclusion Criteria:

* other groups of PH except for CTEPH
* severe renal insufficiency(eGFR<30ml/min·1.73mˆ2)
* severe infectious diseases
* severe hemorrhagic tendency
* severe anaphylaxis of contrast
* pregnancy and lactation
* expected survival time is less than half a year due to tumor or other disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-04-15 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
To evaluate changes of baseline pulmonary vascular resistance (PVR) comparing to that of the final BPA and during follow-up period | at baseline, from enrollment to end of final BPA at 9 months, at 3 months after BPA, at 9 months after BPA, at 15 months after BPA, at 27 months after BPA
  The study will measure pulmonary vascular resistance (PVR) at three time points (baseline before BPA, after final BPA, and follow-up) using right heart catheterization to assess pulmonary hemodynamics by comparing the changes of PVR at above 3 time points.
To evaluate changes of baseline mean pulmonary artery pressure (mPAP) comparing to that of the final BPA and during follow-up period | at baseline, from enrollment to end of final BPA at 9 months, at 3 months after BPA, at 9 months after BPA, at 15 months after BPA, at 27 months after BPA
  The study will measure mean pulmonary artery pressure (mPAP) at three time points (baseline before BPA, after final BPA, and follow-up) using right heart catheterization to assess pulmonary hemodynamics by comparing the changes of mPAP at above 3 time points.

SECONDARY OUTCOMES:
To observe the complications associated with BPA | at baseline, from enrollment to end of final BPA at 9 months, at 3 months after BPA, at 9 months after BPA, at 15 months after BPA, at 27 months after BPA
  The principal complications associated with BPA are pulmonary edema and pulmonary vascular injury, which may lead to symptoms such as hemoptysis, coughing or hypoxia. The study will collect data to assess the incidence of complication and identify risk factor for complications of BPA procedure.
To observe changes of baseline mixed venous oxygen saturation (SvO2) comparing to the final BPA and during follow-up | at baseline, from enrollment to end of final BPA at 9 months, at 3 months after BPA, at 9 months after BPA, at 15 months after BPA, at 27 months after BPA
  Patients with CTEPH commonly manifest hypoxia and decreased exercise capacity due to lower respiratory efficiency. This study will collect oxygen-dynamic data associated with BPA to evaluate respiratory efficiency.
To assess changes of baseline quality of life by calculating SF-36 score comparing to the final BPA and during follow-up | at baseline, from enrollment to end of final BPA at 9 months, at 3 months after BPA, at 9 months after BPA, at 15 months after BPA, at 27 months after BPA
  It has been proved that BPA improve hemodynamic in patients with inoperable CTPEH, but the effect of BPA on QoL has rarely been reported. Each patient will be asked to fill out the SF-36v2 QoL questionnaire before BPA, after final BPA and follow-up period. QoL will be evaluated on 8 scales: physical functioning (PF), role-physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role-emotional (RE) and mental health (MH).Then the investigator will collect 3 time points data to assess changes of QoL in patient with CTEPH.
To evaluate long-term survival after the final BPA procedure and follow-up | at baseline, from enrollment to end of final BPA at 9 months, 1 year postoperative,2 year postoperative
  The primary end point for overall survival analysis is all-cause death. Long-term survival from the initial BPA procedure, the final BPA procedure and follow-up period will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Yuanhua Yang, PhD, Study Chair — Beijing Chao Yang Hospital
Locations (1):
- Beijing Institute of Respiratory Medicine, Beijing Chao-yang Hospital, Capital Medical University, Beijing, China